CLINICAL TRIAL: NCT04257526
Title: Development and Evaluation of a Lifestyle Intervention Among Participants of the French Colorectal Cancer Screening Program
Brief Title: Lifestyle Intervention Among Participants of the French Colorectal Cancer Screening Program
Acronym: LIFE-SCREEN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Centre Leon Berard (Other); Hôpital Edouard Herriot (Other); University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PP201907-26
Record Dates: First submitted 2019-08-30; First posted 2020-02-06 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; prevention
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Colorectal cancer free participants receive evidence-based diet and lifestyle advice in addition to the 'usual care' following a positive FIT test and diagnostic colonoscopy
  Interventions: Behavioral: Diet and lifestyle advice following a positive FIT test and diagnostic colonoscopy.
- Control (No Intervention): Colorectal cancer free participants receive the 'usual care' following a positive FIT test and diagnostic colonoscopy

INTERVENTIONS:
Behavioral: Diet and lifestyle advice following a positive FIT test and diagnostic colonoscopy. — Participants will be recruited during CRC screening and will be included if they have a positive faecal immunochemical test (FIT) and are diagnosed with adenomas but are CRC negative during the colonoscopy. Participants receive evidence-based diet and lifestyle advice intervention with 'usual care'.
  Arms: Intervention

SUMMARY:
The investigators propose a randomized controlled trial to develop and evaluate the impact of promoting advice on diet and lifestyle recommendations for cancer prevention at colorectal cancer screening among individuals who may be at higher risk for colorectal cancer (CRC). The specific objectives of this study are to 1) develop a lifestyle intervention based on evidenced-based diet and lifestyle recommendations (i.e. those proposed by the World Cancer Research Fund (WCRF) and the French National Cancer Institute); 2) evaluate the effect of the intervention on the adherence to the target diet and lifestyle recommendations as well as other subjective health measures, including quality of life; 3) evaluate the effect of the intervention on biological pathways linked to colorectal cancer development including physical fitness, anthropometrics, biomarkers for nutrition, and metabolic health.

DETAILED DESCRIPTION:
This study will be a parallel, two-arm, randomized controlled trial (RCT) in individuals at higher risk of colorectal cancer (CRC), comparing an evidence-based diet and lifestyle advice intervention with 'usual care'. Participants will be recruited during CRC screening and will be included if they have a positive faecal immunochemical test (FIT) and are diagnosed with adenomas but are CRC negative during the colonoscopy. The advice provided will be developed based on the World Cancer Research Fund (WCRF) & French National Cancer Institute (INCA) evidence-based diet and lifestyle recommendations using the habit-theory and will be delivered using multiple materials (e.g. leaflets, posters and digital information) by health professionals in hospitals based in the Rhone region, France. Invitation to participate in the trial will be performed by the gastroenterologist during the clinical visit to provide information on colonoscopy, but the delivery of the intervention and baseline measurement will happen two to three weeks after the colonoscopy. Data will be collected at baseline, 3, 6 and 12 months. At baseline, participants will be required to answer questionnaires on sociodemographic and medical history. At all aforementioned time points, online or paper-based questionnaires will be administered to collect information on diet and lifestyle behaviours, knowledge on healthy lifestyle, quality of life and medical therapy. Participants will also have their anthropometric measures and physical fitness test taken and blood, faecal and colon tissue samples collected during baseline and follow-up appointments (tissue samples will be obtained only for those who are required to undergo the colonoscopy again at 12 months as part of the screening programme). The primary outcome of this intervention will be adherence to target recommendations at 3 months and beyond. Univariate and multivariate statistical analyses as well as qualitative analyses will be performed.

Providing lifestyle advice for cancer prevention at screening programs is a new field in public health that has the potential to be cost-effective, convenient, appealing and wide-reaching. It may also help to reach individuals at higher risk at a time-window when they are more receptive to advice on healthy lifestyles and more likely to make the required behavioural changes. The proposed intervention is expected to have a positive impact on adherence to cancer prevention recommendations, as well as on quality of life, biomarkers for cancer risk, physical fitness and body weight among individuals at higher risk of CRC.

ELIGIBILITY:
Inclusion Criteria:

* At high risk for CRC but CRC negative (confirmed by colonoscopy)
* Able to provide informed consent
* Understanding and able to speak French

Exclusion Criteria:

* Extensive intestinal surgery such as colectomy or surgical resection of the colon
* Chronic gastrointestinal illness (inflammatory bowel disease (IBD), irritable bowel syndrome (IBS), celiac disease)
* Use of any systemic antibiotics, antifungals, antivirals, or antiparasitics in the past 3 months
* Use of probiotic medications in the past 3 months
* Under a strict diet such as meal replacements, diets for co-morbidities such as diabetes
* Immobile due to physical constraints (e.g. handicap that is not compatible with physical activities)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge score assessed via a knowledge questionnaire | 1 year
  The knowledge regarding the effect of lifestyle factors on cancer risk and cancer prevention lifestyle recommendations will be assessed via a knowledge score derived from the General Nutrition & Physical Activity Knowledge Questionnaires
Improvement in lifestyle score assessed via lifestyle questionnaires | 1 year
  WCRF lifestyle score will be assessed through lifestyle questionnaires. Compliance with the WCRF recommendations is considered achieved if this WCRF lifestyle score increases to more than 5 out of 8.
  The following questionnaires will be used to assess lifestyle changes:
  French EPIC food frequency questionnaire; the International Physical Activity Questionnaires - IPAQ; Weight and height measurements to assess BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Marc J Gunter, PhD, Principal Investigator — International Agency for Research on Cancer
Locations (1):
- International Agency for Research on Cancer, Lyon, Rhone, France

IPD SHARING:
Plan to Share IPD: No